CLINICAL TRIAL: NCT00790959
Title: The SASA! Study: a Cluster Randomised Controlled Trial of a Community Mobilisation Intervention to Prevention Violence Against Women and Reduce HIV/AIDS Risk in Kampala, Uganda
Brief Title: The SASA! Study: An Evaluation of a Community Intervention to Address Gender-based Violence and Reduce HIV/AIDS Risk in Uganda
Acronym: SASA!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Raising Voices (Other); Centre for Domestic Violence Prevention, Uganda (Unknown); Makerere University (Other); Sigrid Rausing Trust (Other); Irish Aid (Unknown); Stephen Lewis Foundation (Other)
Responsible Party: Principal Investigator, Charlotte Watts, Professor of Social and Mathematical Epidemiology, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PHHPSASA1
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Intimate Partner Violence; HIV
Keywords: Intimate Partner Violence; HIV/AIDS; Gender; Prevention; Community mobilisation; Uganda
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SASA! (Experimental)
  Interventions: Behavioral: SASA!
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: SASA! — A community mobilization approach to try to change community and individual attitudes and behaviours that support both the perpetration of violence against women and HIV risk behaviours
  The intervention team engages with four major groups of actors: community volunteers selected from the general public; community leaders (e.g. religious, cultural and local council leaders); resource persons (health care providers, police, etc); and institutional leaders. The community volunteers are a key component of the intensive intervention.
  Arms: SASA!
Other: Control — Control communities will receive the full SASA! intervention after completion of the SASA! Study.
  For the duration of the study, they will receive a less intensive intervention comprising the Division-level elements of SASA! (involving community leaders, resource persons and institutional leaders) without the community volunteers.
  Arms: Control

SUMMARY:
The SASA! Study is a cluster randomized trial of a community mobilization intervention for the prevention of HIV and gender based violence. The study is being conducted in Kampala, Uganda.

DETAILED DESCRIPTION:
Background : Physical and sexual violence against women is widespread in Uganda, and is increasingly recognized as a major global social, public health and human rights problem. Epidemiological evidence demonstrates that violence may also be intimately tied in with HIV risk, with violence being both a risk factor for and a consequence of HIV infection.Behaviours that often form the cornerstone of HIV prevention messages such as refusal of sex, inquiring about other partners, or suggesting condom use, have all been identified as triggers of intimate partner violence (IPV) in various settings.

There is now growing interest in integrated HIV/violence prevention strategies to tackle the underlying notions of masculinity that condone both male infidelity and male control over women. Promising research from South Africa and Brazil suggests that interventions which explicitly aim to challenge gender inequalities (either through economic empowerment of women or discussion with men and women about gender inequalities, norms and their implications), may influence levels of violence and HIV risk behaviours. However, such interventions remain few in number, as do scientifically rigorous evaluations of them.

Intervention Design :

SASA! uses a community mobilization approach to address gender inequity and try to change attitudes and behaviours that support both HIV risk behaviours and the perpetration of violence against women.

SASA! supports communities through a four-phase process of social change (based on a social-level adaptation of the Stages of Change Theory):

1. Start to think about violence against women and HIV/AIDS as interconnected issues and the need to personally address these issues
2. Awareness raising about how communities accept men's use of power over women, fueling violence against women and HIV/AIDS
3. Support women and men directly affected by/involved in these issues to change
4. Action to prevent violence against women and HIV/AIDS

The intervention team engages with four major groups of actors: community volunteers selected from the general public; community leaders (e.g. religious, cultural and local council leaders); resource persons (health care providers, police, etc); and institutional leaders. The community volunteers are key agents to raise awareness about power imbalances between men and women, discuss the impacts of HIV and violence against women, discuss the benefits of non-violence and gender equity, and most importantly to mobilize others in the community to take action thereby promoting sustainable change.

Study design:

The SASA! Study randomized four pairs of communities that were matched on population density and stability/transience. The intervention communities received the SASA! intervention from early 2008. Comparison communities will receive the intervention approximately three years later.

A cross-sectional survey will be conducted among community members prior to the implementation of SASA! in their communities. Another cross-sectional survey was initially planned for three years post-implementation, but later delayed to four years post-implementation due to political disturbances that caused interruptions to programme activity. The primary outcomes are: past year experience of physical IPV (among partnered women); past year experience of sexual IPV (among partnered women); acceptability of violence against women; acceptability of a woman refusing sex; community response to women experiencing violence (among women reporting past year physical and/or sexual IPV); and past year concurrent sexual partners (among partnered men). Data analysis will be appropriate to the cluster-randomized study design. The target sample size per arm at each round of data collection is 800.

Complementary qualitative and quantitative data will also be collected (from community volunteers and resource people as well as from community members) to document processes of change and potential pathways of impact.

ELIGIBILITY:
Inclusion Criteria:

* Lived in the community for at least one year
* Aged 18-49 years
* Satisfy gender requirement for sampling sub-cluster

Exclusion Criteria:

* Lack of informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Past year experience of physical violence by an intimate partner (among women partnered in past year) | 4 years after intervention implementation
Past year experience of sexual violence by an intimate partner (among women partnered in the past year) | 4 years after intervention implementation
Acceptability of violence against women | 4 years after intervention implementation
Acceptability of a woman refusing sex | 4 years after intervention implementation
Community response to women experiencing physical and/or sexual IPV in past year (among women reporting physical/sexual IPV in past year) | 4 years after intervention implementation
Past year concurrent sexual partner (among men partnered in past year) | 4 years after intervention implementation

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Watts, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Raising Voices, Kampala, Kampala, Uganda

REFERENCES:
- [Derived] Abramsky T, Musuya T, Namy S, Watts C, Michau L. Changing the norms that drive intimate partner violence: findings from a cluster randomised trial on what predisposes bystanders to take action in Kampala, Uganda. BMJ Glob Health. 2018 Dec 14;3(6):e001109. doi: 10.1136/bmjgh-2018-001109. eCollection 2018. PMID 30613427
- [Derived] Starmann E, Heise L, Kyegombe N, Devries K, Abramsky T, Michau L, Musuya T, Watts C, Collumbien M. Examining diffusion to understand the how of SASA!, a violence against women and HIV prevention intervention in Uganda. BMC Public Health. 2018 May 11;18(1):616. doi: 10.1186/s12889-018-5508-4. PMID 29751754
- [Derived] Abramsky T, Devries KM, Michau L, Nakuti J, Musuya T, Kiss L, Kyegombe N, Watts C. Ecological pathways to prevention: How does the SASA! community mobilisation model work to prevent physical intimate partner violence against women? BMC Public Health. 2016 Apr 16;16:339. doi: 10.1186/s12889-016-3018-9. PMID 27084116
- [Derived] Michaels-Igbokwe C, Abramsky T, Devries K, Michau L, Musuya T, Watts C. Cost and cost-effectiveness analysis of a community mobilisation intervention to reduce intimate partner violence in Kampala, Uganda. BMC Public Health. 2016 Feb 29;16:196. doi: 10.1186/s12889-016-2883-6. PMID 26924488
- [Derived] Abramsky T, Devries KM, Michau L, Nakuti J, Musuya T, Kyegombe N, Watts C. The impact of SASA!, a community mobilisation intervention, on women's experiences of intimate partner violence: secondary findings from a cluster randomised trial in Kampala, Uganda. J Epidemiol Community Health. 2016 Aug;70(8):818-25. doi: 10.1136/jech-2015-206665. Epub 2016 Feb 12. PMID 26873948
- [Derived] Kyegombe N, Abramsky T, Devries KM, Starmann E, Michau L, Nakuti J, Musuya T, Heise L, Watts C. The impact of SASA!, a community mobilization intervention, on reported HIV-related risk behaviours and relationship dynamics in Kampala, Uganda. J Int AIDS Soc. 2014 Nov 5;17(1):19232. doi: 10.7448/IAS.17.1.19232. eCollection 2014. PMID 25377588
- [Derived] Abramsky T, Devries K, Kiss L, Nakuti J, Kyegombe N, Starmann E, Cundill B, Francisco L, Kaye D, Musuya T, Michau L, Watts C. Findings from the SASA! Study: a cluster randomized controlled trial to assess the impact of a community mobilization intervention to prevent violence against women and reduce HIV risk in Kampala, Uganda. BMC Med. 2014 Jul 31;12:122. doi: 10.1186/s12916-014-0122-5. PMID 25248996
- [Derived] Abramsky T, Devries K, Kiss L, Francisco L, Nakuti J, Musuya T, Kyegombe N, Starmann E, Kaye D, Michau L, Watts C. A community mobilisation intervention to prevent violence against women and reduce HIV/AIDS risk in Kampala, Uganda (the SASA! Study): study protocol for a cluster randomised controlled trial. Trials. 2012 Jun 29;13:96. doi: 10.1186/1745-6215-13-96. PMID 22747846